CLINICAL TRIAL: NCT05948462
Title: Phase II Study of Lorlatinib in Combination With Chemotherapy in Participants With Metastatic Anaplastic Lymphoma Kinase Positive (ALK+) Non-small Cell Lung Cancer (NSCLC) Who Progressed on Single-agent Lorlatinib
Brief Title: Lorlatinib in Combination With Chemotherapy in Participants With Metastatic Anaplastic Lymphoma Kinase Positive (ALK+) Non-small Cell Lung Cancer (NSCLC) Who Progressed on Single-agent Lorlatinib
Acronym: NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn by pharmaceutical funding partner
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN 481
Record Dates: First submitted 2023-06-27; First posted 2023-07-17 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: ALK positive; ALK+; Metastatic; Lung; NSCLC; Non-small cell lung cancer; Lorlatinib; Small molecule kinase inhibitor; Pemetrexed; Carboplatin; Cisplatin
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — lorlatinib; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lorlatinib and Platinum and Pemetrexed (Experimental): Lorlatinib will be administered by mouth daily plus Pemetrexed by IV infusion every 3 weeks until progression or intolerable toxicity. Platinum-based standard of care chemotherapy by IV infusion will also be given every 3 weeks for the first 4 cycles; carboplatin or cisplatin are the platinum agents that may be selected based on physician discretion. One cycle is defined as 3 weeks.
  Interventions: Drug: Lorlatinib; Drug: Cisplatin or Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Lorlatinib — Participants will receive assigned dose of daily oral lorlatinib continuously for each cycle. Each cycle is 3 weeks.
  Other Names: Lorbrena; Lorviqua
Drug: Cisplatin or Carboplatin — Participants will receive standard of care intravenous Cisplatin or Carboplatin, both chemotherapy medications, on day 1 of each cycle every 3 weeks, for Cycles 1-4. Each cycle is 3 weeks.
  Other Names: Platinol (Cisplatin); Paraplatin (Carboplatin)
Drug: Pemetrexed — Participants will receive intravenous Pemetrexed, a chemotherapy medication, on day 1 of each cycle. Each cycle is 3 weeks.
  Other Names: Alimta; Pemfexy; Ciambra

SUMMARY:
This clinical trial is an open-label, single arm study evaluating the safest dose of lorlatinib in combination with standard of care chemotherapy in participants with metastatic anaplastic lymphoma kinase positive (ALK+) NSCLC who progressed on prior therapy of lorlatinib alone. The main goals of this study are to:

* Evaluate the safety and tolerability of lorlatinib in combination with standard of care chemotherapy.
* Evaluate how well the combination of lorlatinib and standard of care chemotherapy works to treat metastatic anaplastic lymphoma kinase positive (ALK+) NSCLC.
* Evaluate the pharmacokinetics (PK) of lorlatinib when given in combination with standard of care chemotherapy.

DETAILED DESCRIPTION:
Lorlatinib is a kinase inhibitor with in vitro activity against ALK and ROS1. This study's aim is to evaluate the safety of lorlatinib given in combination with platinum-based standard of care chemotherapy in participants with metastatic anaplastic lymphoma kinase positive (ALK+) non-small-cell lung cancer who progressed after receiving lorlatinib alone.

There will be a lead-in portion for the first six participants treated. Lead-in participants will receive an assigned starting dose of lorlatinib by mouth once daily throughout each cycle. In addition, a platinum-based standard of care chemotherapy regimen, to include carboplatin or cisplatin as well as pemetrexed, will be given intravenously every 3 weeks. A cycle is defined as 3 weeks. After tolerability is confirmed in the lead-in with the first 6 participants on trial, the next 9 participants may begin at an increased starting dose of lorlatinib by mouth once daily. After 4 cycles of oral lorlatinib and intravenous platinum-based standard of care chemotherapy and intravenous pemetrexed, the participant will move into the maintenance regimen. The maintenance regimen will include continuing on daily oral lorlatinib plus intravenous pemetrexed every 3 weeks until disease progression or intolerable toxicity or other reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, according to local guidelines, signed and dated by the participant or by a legal guardian prior to the performance of any study-specific procedures, sampling, or analyses
2. At least 18 years-of-age at the time of signature of the informed consent form (ICF)
3. Metastatic ALK+ NSCLC
4. Clinical and/or radiological progressive disease while receiving lorlatinib monotherapy or within 3 weeks of stopping lorlatinib monotherapy due to clinical and/or radiological progressive disease
5. Adequate hematologic function defined as:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Hemoglobin (Hb) ≥9 g/dL
   * Platelets ≥100,000/μL
6. Adequate liver function defined as:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × the upper limit of normal (ULN)
   * Total bilirubin ≤1.5 × ULN (Participants with known Gilbert disease: serum bilirubin level ≤ 3 × ULN)
7. Adequate renal function defined as calculated creatinine clearance ≥45 mL/min as calculated by Cockcroft and Gault Formula
8. Male or female participants. Male participants with female partners of childbearing potential and female participants of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 90 days following last dose. Male participants must also refrain from donating sperm during their participation in the study.

Exclusion Criteria:

1. Prior treatment with platinum-based standard of care doublet chemotherapy with pemetrexed
2. ECOG Performance Status score ≥3
3. Current treatment with any of the following:

   * Known strong CYP3A inhibitors (e.g., atazanavir, boceprevir, clarithromycin, conivaptan, indinavir, itraconazole, ketoconazole, lopinavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, troleandomycin, voriconazole, grapefruit juice or grapefruit/grapefruit-related citrus fruits [e.g., Seville oranges, pomelos]). The topical use of these medications (if applicable), such as 2% ketoconazole cream, is allowed.
   * Known strong CYP3A inducers (e.g., avasimibe, carbamazepine, phenobarbital, phenytoin, rifatutin, rifampin, St. John's Wort)
   * CYP3A substrates with a narrow therapeutic index (e.g., alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl including transdermal patch, pimozide, quinidine, sirolimus, tacrolimus) within 12 days prior to the first dose of lorlatinib
   * Known P-gp substrates with a narrow therapeutic index (e.g., digoxin)
   * Currently receiving treatment with therapeutic doses of warfarin sodium. Low- molecular-weight heparin is allowed.
   * Major surgery (excluding placement of vascular access) within 4 weeks of first dose of study drug(s).
4. Has any history of ILD (including pulmonary fibrosis or radiation pneumonitis), has clinically significant ILD, or is suspected to have such disease by imaging during screening. If imaging findings are unlikely to indicate a history of pneumonitis, then the Investigator should discuss the considerations with the Study Chair about potential enrollment and record the reasoning in the source documentation.
5. Clinically severe pulmonary compromise (based on Investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

   * any underlying pulmonary disorder (e.g., severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease)
   * any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (e.g., rheumatoid arthritis, Sjögren's syndrome, sarcoidosis) OR prior pneumonectomy
6. Women who are pregnant, nursing, or plan to become pregnant while in the study and for at least 6 months after the last administration of study treatment
7. Men who plan to father a child while in the study and for at least 3 months after the last administration of study treatment
8. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of lorlatinib (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2, malabsorption syndrome)
9. Any of the following cardiac criteria:

   * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting electrocardiograms (ECGs), e.g., complete left bundle branch block, third-degree heart block
   * Congestive heart failure (New York Heart Association ≥ Grade 2)
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval
   * Second degree or third-degree AV block (unless paced) or any AV block with PR >220 msec
10. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection, including hepatitis B, hepatitis C, and human immunodeficiency virus. Screening for chronic conditions is not required.
11. Presence of other active invasive cancers other than the one treated in this study within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse and serious adverse events of lorlatinib in combination with standard of care platinum-based chemotherapy and pemetrexed as assessed by CTCAE v5.0. | From Cycle 1 Day 1 to 30 days after treatment discontinuation, up to approximately 1 year. Each cycle is 3 weeks.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) analysis: lowest concentration with steady state dosing interval (Css, min) of lorlatinib in combination with standard of care platinum-based chemotherapy and pemetrexed. | Cycle 1, Day 1; Cycle 2, Day 1; Cycle 4, Day 1 (each cycle is 3 weeks) and at time of treatment discontinuation, up to approximately 1 year.
Objective Response Rate (ORR) to assess the anti-tumor activity of treatment with lorlatinib in combination with standard of care platinum-based chemotherapy and pemetrexed. | Up to approximately 26 months
  Percentage of participants demonstrating a Complete Response (CR) or Partial Response (PR) according to RECIST v1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, MD, Study Chair — SCRI Development Innovations, LLC
Locations (5):
- United States (5):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Messino Cancer Center, Asheville, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No